CLINICAL TRIAL: NCT04446182
Title: A Phase II Study of Itacitinib (INCB039110) and Extracorporeal Photopheresis (ECP) for First-Line Treatment in Chronic Graft Versus Host Disease (GVHD)
Brief Title: Itacitinib (INCB039110) and Extracorporeal Photopheresis (ECP) for First-Line Treatment in Chronic GVHD
Acronym: FLIGHT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Utah (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI130090
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Chronic Graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — itacitinib; INCB039110; Photopheresis

STUDY DESIGN:
Intervention Model Description: The RP2D will be determined by a 3+3 dose de-escalation design. Once an RP2D has been confirmed, Part 2 will open as an expansion cohort. (As this study was terminated after enrolling 3 patients, Part 2 of the planned study did not occur.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental): Patients will self-administer itacitinib every morning regardless of food. ECP will be administered twice weekly on consecutive days for 8 weeks per institutional standards. At the end of 8 weeks of combination therapy, patients will start a standard ECP taper schedule and itacitinib will be continued at the assigned dose level. After six cycles of therapy, itacitinib may be tapered at the treating investigator's discretion as described below.
  Interventions: Drug: Itacitinib; Device: Extracorporeal Photopheresis (ECP)

INTERVENTIONS:
Drug: Itacitinib — All eligible patients will begin study therapy with approximately a week lead-in of itacitinib monotherapy at scheduled dose. Itacitinib will be taken daily at scheduled dose for a total of six cycles. Itacitinib may be tapered as deemed appropriate by the treating investigator. Patients will remain on study therapy as long as treatment discontinuation criteria are not met. Patients with Partial Response (PR) or better may continue itacitinib for up to 1 year.
  Other Names: INCB039110
Device: Extracorporeal Photopheresis (ECP) — ECP will begin after itacitinib lead in period. At the end of 8 weeks of combination therapy, patients will start a standard ECP taper schedule. Patients achieving PR or better after 6 cycles of itacitinib may continue treatment with itacitinib for up to 1 year. Thereafter, itacitinib may be tapered at the treating investigator's discretion.
  Other Names: ECP

SUMMARY:
An open-label, Phase II trial designed to assess the recommended phase 2 dose (RP2D) of itacitinib in combination ECP and efficacy of the combination after 24 weeks of therapy. The trial will consist of two parts: Part One will assess the RP2D. For dose-finding purposes, the dose limiting toxicity (DLT) evaluation period will be defined as the time from the first dose of itacitinib lead-in (7-day lead-in) to the last day of cycle one combination therapy (Cycle one day 28).

Part Two will further describe and characterize the safety and efficacy of the regimen. The RP2D will be determined by a 3+3 dose de-escalation design. Should dose level one be deemed intolerable, enrollment will proceed at dose level -1. The RP2D will be affirmed according to the rules of the 3+3 dose de-escalation scheme. Once an RP2D has been confirmed, Part 2 will open as an expansion cohort.

As this study was terminated after enrolling three patients out of an anticipated target accrual of 58, Part Two of this study did not occur.

ELIGIBILITY:
Inclusion Criteria:

* -Male or female subject aged ≥ 18 years.
* Active, clinically diagnosed, moderate or severe chronic GVHD as defined by the NIH Consensus Development Project Criteria (See Appendix 2).
* History of an allogeneic hematopoietic cell transplant with any conditioning regimen, donor, or graft source.
* Need for systemic treatment for chronic GVHD as assessed by the treating investigator.
* No previous systemic treatment for chronic GVHD. Note: Participants may be receiving immunosuppressants for the prophylaxis or treatment of acute GVHD, but these medications must have been stable for at least 2 weeks prior to the initiation of study therapy. Prednisone dose (or its equivalent) should be at doses of ≤0.25 mg/kg/d for at least 2 weeks prior to the initiation of study therapy.

Topical or inhaled treatments for chronic GVHD are allowed. Any prior ECP treatments for the management of acute GVHD must have occurred > 4 weeks prior to the initiation of itacitinib treatment.

* Able to swallow and retain oral medication.
* Life expectancy > 24 weeks.
* Karnofsky performance status ≥ 60
* Evidence of myeloid and platelet engraftment:

  * Absolute neutrophil count ≥ 1000/microliter (mcL)
  * Platelet count ≥ 25,000/mcL

Note: Use of growth factors and transfusion support is allowed during the study; however, growth factors and transfusion support to reach a minimum absolute neutrophil count (ANC) or platelet count for inclusion are not allowed within the 7 days before the screening laboratory assessment.

* Adequate organ function as defined as:

  * Hepatic:

    * Total bilirubin ≤ 2 mg/dL
    * alanine transaminase (AST)(SGOT)/aspartate aminotransferase (ALT)(SGPT) ≤ 2.5 × institutional upper limit of normal (ULN) (unless of non-hepatic origin). AST/ALT ≤ 5 x ULN is acceptable if associated with chronic GVHD.
  * Renal:

    ---estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 as calculated using the Modification of Diet in Renal Disease formula or by the Cockcroft-Gault formula:
    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
    * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
  * Coagulation:

    * PT/ international normalized ratio (INR) < 1.5 x ULN and PTT (aPTT) < 1.5 x ULN (unless abnormalities are unrelated to coagulopathy or bleeding disorder). When treated with warfarin or other vitamin K antagonist, then INR ≤ 3 x ULN.
* Willingness to avoid pregnancy or father children based on the criteria below and as described in Section 5.4.2:

  * Woman of non-childbearing potential (i.e., surgically sterile with a hysterectomy and/or bilateral oophorectomy for at least 3 months OR ≥ 12 months of amenorrhea and at least 50 years of age).
  * Woman of childbearing potential who has a negative serum pregnancy test at screening and negative urinary test before the first dose on Day 1 and who agrees to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the subject and their understanding confirmed.
  * Men who agree to take appropriate precautions to avoid fathering children (with at least 99% certainty) from screening through safety follow-up. Permitted methods that are at least 99% effective in preventing pregnancy should be communicated to the subject and their understanding confirmed.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Subjects with score 3 lung GVHD; or biopsy-proven bronchiolitis obliterans.
* Participants have uncontrolled manifestations of acute GVHD.
* Treatment with any investigational medication within ≤ 30 days or 5 half-lives, whichever is longer, before the first dose of study drug.
* Patients who have received any previous systemic treatment for chronic GVHD, including corticosteroids, prior to Cycle 1, Day 1.

Note: Prior and concomitant use of Calcineurin-Inhibitors (CNIs) for prevention and treatment of acute GVHD, as well as topical/inhaled steroids, is acceptable.

* Received prior Janus kinase (JAK) inhibitor therapy for any indication ≤ 4 weeks prior to Cycle 1 Day 1.
* Patients with relapsed or progressive malignant disease or any post-transplant lymphoproliferative disease.
* Chronic GVHD occurring after a non-scheduled donor lymphocyte infusion (DLI) administered for pre-emptive treatment of malignancy recurrence. Participants who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes the administration of oral medications.
* Any contraindication for extracorporeal photopheresis (ECP) per the treating investigator's discretion.
* Subject has a concurrent illness which in the opinion of the investigator may interfere with the treatment and evaluation of the subject.
* Pregnant or currently breast-feeding. Note: INCB039110 is a Janus kinase 1 (JAK1) inhibitor with the potential for serious or life-threatening birth defects or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with INCB039110, breastfeeding should be discontinued if the mother is treated with INCB039110. These potential risks may also apply to other agents used in this study.
* Vaccinated with live, attenuated vaccines within 4 weeks of the first dose of study drug and while on trial.
* Use of any prohibited concomitant medications as described in Section 6.5. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment.
* Inadequate recovery from toxicity and/or complications from major surgery before starting therapy.
* Unwillingness to be transfused with blood components during the study.
* History of other malignancy (not including the underlying malignancy that was the indication for the transplant), with the following exceptions:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to Screening and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease.
  * Adequately treated cervical carcinoma in situ without current evidence of disease.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months of enrollment, New York Heart Association (NYHA) Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or an arrhythmia that requires therapy.
  * A clinically significant respiratory disease that requires mechanical ventilation support or ≥ 50% oxygen.
  * Any uncontrolled active systemic infection or active infection requiring systemic treatment that was ongoing ≤ 7 days before screening. Subjects with acute infections requiring treatment should delay screening/enrollment until the course of therapy has been completed and the event is considered resolved. Prophylactic antibiotics will be permitted.
  * Cholestatic disorders, or unresolved sinusoidal obstructive syndrome/ veno-occlusive disease of the liver (defined as persistent total bilirubin > 2 mg/dL, or abnormalities not attributable to GVHD and ongoing organ dysfunction).
* History of thromboembolic event within 1 month before study registration.
* HIV-infected patients on effective antiretroviral therapy with an undetectable viral load within 6 months are eligible for this trial.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection that requires treatment, or at risk for HBV reactivation (i.e., positive HBsAg). Participants with negative HBsAg and positive total hepatitis B core antigen (HBc) antibody may be included if HBV DNA is undetectable at the time of screening. Participants who are positive for HCV antibodies are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA. Participants whose immune status is unknown or uncertain must have results confirming immune status before enrollment. Serology results performed less than or equal to 6 months prior to the first planned dose of itacitinib are acceptable for determining eligibility.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug/treatment and attending required study visits; pose a significant risk to the participant; or interfere with the interpretation of study data.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations) per the investigator's assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lee, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: All Participants (Dose Level 1, Starting Dose): Participants will begin with a 5-10 lead-in period of self-administered itacitinib, after which they will continue itacitinib for 6 28 day cycles. Extracorporeal Photopheresis (ECP) will begin on Cycle 1 Day 1 after the lead-in period, and will be administered twice weekly on consecutive days for 8 weeks. At the end of 8 weeks (2 cycles) of combination therapy, participants will start a standard ECP taper schedule and itacitinib will be continued at the assigned dose level. After six cycles of therapy, itacitinib may be tapered at the treating investigator's discretion.
  Though this study was initially conceived as a dose de-escalation study, the study was terminated with three participants accrued, meaning all patients received the starting dose of 200 mg daily, days 1-28 per cycle, per the 3+3 dose de-escalation study design. Thus, only one treatment arm is appropriate in reporting study results.
Period: Overall Study
Arm/Group | Treatment: All Participants (Dose Level 1, Starting Dose)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: All Participants: Participants will begin with a 5-10 lead-in period of self-administered itacitinib, after which they will continue itacitinib for 6 28 day cycles. Extracorporeal Photopheresis (ECP) will begin on Cycle 1 Day 1 after the lead-in period, and will be administered twice weekly on consecutive days for 8 weeks. At the end of 8 weeks (2 cycles) of combination therapy, participants will start a standard ECP taper schedule and itacitinib will be continued at the assigned dose level. After six cycles of therapy, itacitinib may be tapered at the treating investigator's discretion.
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.33 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
Mean Baseline NIH Global GVHD Score [Mean (Standard Deviation); unit: score on a scale] — Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline. This data point in the criteria is an overall global rating of the participant's GVHD, ranging from 0 (no GVHD) to 3 (severe GVHD).
  score on a scale | 2 (0)
Mean clinician-assessed NIH GVHD severity score [Mean (Standard Deviation); unit: score on a scale] — Participants were assessed by the treating clinician for chronic graft versus host disease (cGVHD) symptom severity per the NIH Consensus Development Project Criteria at baseline. One data point in the criteria is a general rating the severity of the participant's GVHD symptoms, ranging from 0 (GVHD symptoms not at all severe) to 10 (most severe GVHD symptoms possible).
  score on a scale | 4.67 (.58)
Mean participant-assessed NIH GVHD severity score [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to rate their own symptoms for chronic graft versus host disease (cGVHD) severity per the NIH Consensus Development Project Criteria at baseline. One data point in is a general rating of the severity of the participant's GVHD symptoms, ranging from 0 (GVHD symptoms not at all severe) to 10 (most severe GVHD symptoms possible).
  score on a scale | 6.33 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With a Dose-limiting Toxicity (DLT) During the DLT Evaluation Period.
Description: Adverse events were assessed at each study visit from the first dose of itacitinib during the lead-in period (lead-in period = 5-10 days) until the last day of cycle one (each cycle = 28 days) of combination treatment with itacitinib and Extracorporeal Photopheresis (ECP). A DLT was defined as an Adverse Event (AE) that was 1) attributed as possibly, probably, or definitely related to itacitinib or to the combination of itacitinib and ECP, and 2) graded as "severe" or "life threatening" (grade 3 or 4) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Time Frame: up to 38 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Count of Participants With a Response to Treatment at 24 Weeks of Treatment
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline and after 24 weeks of treatment. The criteria evaluates 9 organ systems, and then defines a partial response (PR) as at least one organ system with improvement since baseline and no worsening in other organs. Complete response (CR) is defined as an improvement in all affected organ systems to having no GVHD symptoms in any organ system. All responses must occur without any secondary systemic immunosuppressive therapy, and no malignancy recurrence or death. Participants with a PR or CR are counted as a response for this outcome.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: Count of Participants Who Experience Adverse Events (AEs) and Serious Adverse Events (SAEs) During Study Treatment
Description: Adverse events were assessed at each study visit per CTCAE v5 criteria. This objective counts the number of participants who experienced 1) any adverse event of any severity, or 2) any serious adverse event that was possibly, probably, or definitely related to itacitinib or to combination treatment with itacitinib and ECP.
Time Frame: during study treatment - up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants
  Adverse Events | 3
  Serious Adverse Events | 1

4. Secondary Outcome: Count of Participants With a Response to Treatment After One Year of Treatment
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline and after one year of treatment. The criteria evaluates 9 organ systems, and then defines a partial response (PR) as at least one organ system with improvement since baseline and no worsening in other organs. Complete response (CR) is defined as an improvement in all affected organ systems to having no GVHD symptoms in any organ system. All responses must occur without any secondary systemic immunosuppressive therapy, and no malignancy recurrence or death. Participants with a PR or CR are counted as a response for this outcome.
Time Frame: 1 year
Population: Only one participant was assessed at the one year time point. The others had discontinued treatment prior to that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Count of Participants With Failure Free Survival (FFS) at 24 Weeks and 1 Year
Description: Failure Free Survival (FFS) is defined as the number of participants at 24 weeks and at 1 year who have not experienced treatment failure. Treatment failure is defined as the initiation of secondary therapy for chronic GVHD, malignancy relapse, or death from any cause.
Time Frame: 24 weeks and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants
  FFS at 24 weeks | 3
  FFS at 1 year | 2

6. Secondary Outcome: Count of Participants Who Have Withdrawn All Immunosuppressants at 1 Year
Description: Immunosuppressive therapy is common for participants with GVHD. This objective counts the number of participants who were able to discontinue all immunosuppressants by 1 year of treatment and follow-up.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants | 0

7. Secondary Outcome: Count of Participants With a Response to Treatment at 24 Weeks of Treatment Stratified by Concurrent Prednisone Use
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline and after 24 weeks of treatment. The criteria evaluates 9 organ systems, and then defines a partial response (PR) as at least one organ system with improvement since baseline and no worsening in other organs. Complete response (CR) is defined as an improvement in all affected organ systems to having no GVHD symptoms in any organ system. All responses must occur without any secondary systemic immunosuppressive therapy, and no malignancy recurrence or death. Participants with a PR or CR are counted as a response for this outcome. Participants were also evaluated for the amount of prednisone (or other steroids converted by prednisone equivalence) they were using at the time of the response. This outcome is the same as outcome # 2, but has been stratified by prednisone use.
Time Frame: 24 weeks
Population: Two participants, both at the 0 mg/kg/d prednisone use, were assessed for this measure at 24 weeks. The other had discontinued treatment prior to that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 2
Participants
  0 mg/kg/d prednisone use | 2
  ≤ 0.25mg/kg/d prednisone use: number analyzed (Participants) | 0
  ≤ 0.25mg/kg/d prednisone use | 0
  > 0.25mg/kg/d prednisone use: number analyzed (Participants) | 0
  > 0.25mg/kg/d prednisone use | 0

8. Secondary Outcome: Mean Cumulative Prednisone Used up to 24 Weeks
Description: This outcome assessed the cumulative amount of prednisone (or other steroids converted to prednisone equivalence) used by participants up to 24 weeks of treatment.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
milligrams | 30 (42.426)

9. Secondary Outcome: Count of Participants With Organ-specific Responses at 24 Weeks
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline and after 24 weeks of treatment. The criteria evaluate 9 organ systems, and for each organ, defines changes in symptoms to qualify as a partial response (PR), complete response (CR), or progressive disease (PD) in that organ. In general, PR in an organ indicates partial improvement after prior involvement of that organ. CR indicates improvement to no symptoms after prior involvement. PD indicates worsening of symptoms in the organ system. Lack of response indicates that the organ system was involved at both baseline and 24 weeks, but did not improve or deteriorate sufficiently to qualify for PR, CR, or PD. No involvement/Not evaluable indicates that the organ system never had any GVHD symptoms or was not able to be evaluated.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants
  Mouth: Progression | 0
  Mouth: Partial Response | 0
  Mouth: Complete Response | 3
  Mouth: Lack of response | 0
  Mouth: No involvement/Not evaluable | 0
  Eyes: Progression | 0
  Eyes: Partial Response | 0
  Eyes: Complete Response | 1
  Eyes: Lack of response | 0
  Eyes: No involvement/Not evaluable | 2
  Skin: Progression | 0
  Skin: Partial Response | 2
  Skin: Complete Response | 0
  Skin: Lack of response | 1
  Skin: No involvement/Not evaluable | 0
  Esophagus: Progression | 0
  Esophagus: Partial Response | 0
  Esophagus: Complete Response | 0
  Esophagus: Lack of response | 0
  Esophagus: No involvement/Not evaluable | 3
  Upper GI: Progression | 0
  Upper GI: Partial Response | 0
  Upper GI: Complete Response | 0
  Upper GI: Lack of response | 0
  Upper GI: No involvement/Not evaluable | 3
  Lower GI: Progression | 0
  Lower GI: Partial Response | 0
  Lower GI: Complete Response | 0
  Lower GI: Lack of response | 0
  Lower GI: No involvement/Not evaluable | 3
  Liver: Progression | 0
  Liver: Partial Response | 0
  Liver: Complete Response | 0
  Liver: Lack of response | 0
  Liver: No involvement/Not evaluable | 3
  Lungs: Progression | 0
  Lungs: Partial Response | 0
  Lungs: Complete Response | 0
  Lungs: Lack of response | 0
  Lungs: No involvement/Not evaluable | 3
  Joints and facia: Progression | 1
  Joints and facia: Partial Response | 2
  Joints and facia: Complete Response | 0
  Joints and facia: Lack of response | 0
  Joints and facia: No involvement/Not evaluable | 0

10. Secondary Outcome: Count of Participants With Organ-specific Responses at 1 Year
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline and after 1 year of treatment. The criteria evaluate 9 organ systems, and for each organ, defines changes in symptoms to qualify as a partial response (PR), complete response (CR), or progressive disease (PD) in that organ. In general, PR in an organ indicates partial improvement after prior involvement of that organ. CR indicates improvement to no symptoms after prior involvement. PD indicates worsening of symptoms in the organ system. Lack of response indicates that the organ system was involved at both baseline and 24 weeks, but did not improve or deteriorate sufficiently to qualify for PR, CR, or PD. No involvement indicates that the organ system never had any GVHD symptoms.
Time Frame: 1 year
Population: Only one participant completed 1 year of treatment to be evaluated for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 1
Participants
  Mouth: Progression | 0
  Mouth: Partial Response | 1
  Mouth: Complete Response | 0
  Mouth: Lack of Response | 0
  Mouth: No involvement/Not evaluable | 0
  Eyes: Progression | 1
  Eyes: Partial Response | 0
  Eyes: Complete Response | 0
  Eyes: Lack of Response | 0
  Eyes: No involvement/Not evaluable | 0
  Skin: Progression | 0
  Skin: Partial Response | 1
  Skin: Complete Response | 0
  Skin: Lack of Response | 0
  Skin: No involvement/Not evaluable | 0
  Esophagus: Progression | 0
  Esophagus: Partial Response | 0
  Esophagus: Complete Response | 0
  Esophagus: Lack of Response | 0
  Esophagus: No involvement/Not evaluable | 1
  Upper GI: Progression | 0
  Upper GI: Partial Response | 0
  Upper GI: Complete Response | 0
  Upper GI: Lack of Response | 0
  Upper GI: No involvement/Not evaluable | 1
  Lower GI: Progression | 0
  Lower GI: Partial Response | 0
  Lower GI: Complete Response | 0
  Lower GI: Lack of Response | 0
  Lower GI: No involvement/Not evaluable | 1
  Liver: Progression | 0
  Liver: Partial Response | 0
  Liver: Complete Response | 0
  Liver: Lack of Response | 0
  Liver: No involvement/Not evaluable | 1
  Lungs: Progression | 0
  Lungs: Partial Response | 0
  Lungs: Complete Response | 0
  Lungs: Lack of Response | 0
  Lungs: No involvement/Not evaluable | 1
  Joints and facia: Progression | 0
  Joints and facia: Partial Response | 0
  Joints and facia: Complete Response | 1
  Joints and facia: Lack of Response | 0
  Joints and facia: No involvement/Not evaluable | 0

11. Secondary Outcome: Mean NIH Global GVHD Score at 24 Weeks
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline and after 24 weeks of treatment. One data point in the criteria is an overall global rating of the participant's GVHD, ranging from 0 (no GVHD) to 3 (severe GVHD). The baseline global score is reported in the baseline characteristics.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
score on a scale | 1.67 (.58)

12. Secondary Outcome: Duration of Response (DOR)
Description: DOR was measured as the interval between the date of initial documentation of a response (PR or better), and the date of progression, start of a new therapy for chronic GVHD (cGVHD) (including corticosteroids), or death from any cause.
Time Frame: up to 1 year
Population: Two participants had a partial response or better.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 2
days | 119.5 (93.5)

13. Secondary Outcome: Mean Clinician-evaluated GVHD Severity Score at 24 Weeks and 1 Year
Description: Participants were assessed for chronic graft versus host disease (GVHD) severity per the NIH Consensus Development Project Criteria at baseline, after 24 weeks of treatment, and after one year of treatment. One data point in the criteria is a general rating the severity of the participant's GVHD symptoms, ranging from 0 (GVHD symptoms not at all severe) to 10 (most severe GVHD symptoms possible). The baseline severity score is reported in the baseline characteristics.
Time Frame: at 24 weeks and 1 year
Population: Only one participant continued treatment long enough to be evaluated at 1 year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
score on a scale
  Severity score at 24 weeks | 4 (1.73)
  Severity score at 1 year: number analyzed (Participants) | 1
  Severity score at 1 year | 3 (0)

14. Secondary Outcome: Mean Participant-reported cGVHD Symptom Severity Score at 24 Weeks and at 1 Year
Description: Participants were asked to rate their own symptoms for chronic graft versus host disease (cGVHD) severity per the NIH Consensus Development Project Criteria at baseline, after 24 weeks of treatment, and after one year of treatment. One data point in is a general rating of the severity of the participant's GVHD symptoms, ranging from 0 (GVHD symptoms not at all severe) to 10 (most severe GVHD symptoms possible). The baseline severity score is reported in the baseline characteristics.
Time Frame: 24 weeks and 1 year
Population: One participant did not complete the cGVHD severity assessment at week 24. Two participants did not continue treatment long enough to self-assess for cGVHD severity at one year.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 2
score on a scale
  Severity score at 24 weeks | 6 (1.41)
  Severity score at 1 year: number analyzed (Participants) | 1
  Severity score at 1 year | 5 (0)

15. Secondary Outcome: Count of Participants With Non-relapse Mortality (NRM)
Description: NRM is defined as death due to causes other than a relapse of their primary hematologic disease. This outcome reports the number of participants who were deceased at 24 weeks and at 1 year after the start of treatment whose death meets the definition of NRM.
Time Frame: 24 weeks and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants
  NRM at 24 weeks | 0
  NRM at 1 year | 0

16. Secondary Outcome: Count of Participants With Relapse at 24 Weeks and 1 Year
Description: Relapse is defined as re-activation of the participant's primary hematologic malignancy after it has been in remission. This outcome reports the number of participants who had experienced relapse at 24 weeks and at 1 year after start of treatment.
Time Frame: 24 weeks and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants
  Relapse at 24 weeks | 0
  Relapse at 1 year | 0

17. Secondary Outcome: Count of Participants Alive at 24 Weeks and 1 Year
Description: This outcome measures overall survival (OS), meaning the number of participants who remain alive at 24 weeks and at 1 year from start of treatment.
Time Frame: 24 weeks and 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment: All Participants
Number analyzed (Participants) | 3
Participants
  Overall Survival at 24 weeks | 3
  Overall Survival at 1 year | 3

ADVERSE EVENTS:
Time Frame: Collection of serious adverse events will begin at the initiation of study treatment and end 30 days after the last dose of study treatment or until new cancer treatment is initiated, whichever happens the soonest. For this study, actual treatment ranged from 181 days to 350 days with a median of 203 days.
Description: Adverse events were reviewed with the participant and the investigator at every study visit. All adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, were collected.
Arm/Group | Treatment: All Participants
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment: All Participants (N=3)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — human metapneumovirus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment: All Participants (N=3)
Dry eye (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1/2 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (6)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT04446182/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT04446182/ICF_001.pdf